CLINICAL TRIAL: NCT02309164
Title: The Use of Acupuncture for Treatment of Chemotherapy-induced Peripheral Neuropathy (CIPN).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rebeca Boltes Cecatto, Rebeca Boltes Cecatto, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 261/14
Record Dates: First submitted 2014-09-16; First posted 2014-12-05 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Neoplasm; Adult Disease; Neuropathy
MeSH Terms: conditions — Neoplasms; Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Active Comparator): acupuncture
  Interventions: Procedure: Acupuncture; Behavioral: Orientation group
- orientation group (Sham Comparator): medical management guidelines for foot / hands care, sensory desensitization, risk prevention guidelines, proper ergonomics and orthoses when necessary.
  Interventions: Behavioral: Orientation group

INTERVENTIONS:
Procedure: Acupuncture — 10 acupuncture sessions of 30 minutes each, twice a week
  Arms: Acupuncture
Behavioral: Orientation group — medical management guidelines for foot / hands care, sensory desensitization, risk prevention guidelines, proper ergonomics and orthoses when necessary.

SUMMARY:
This study aims to determine the effectiveness of the use of acupuncture in relieving sensory and motor symptoms as well as functional impairment and quality of life of patients with chemotherapy induced peripheral neuropathy

DETAILED DESCRIPTION:
The trial is a clinical, single-center, randomized trial study that will involve 30 adult cancer patients with chemotherapy-induced peripheral neuropathy randomized into two groups (control and acupuncture treated with 10 sessions, 2X per week). Both CIPN patients groups will be submitted to a complete physical examination and to clinical assessments with National Cancer Institute Common Terminology Criteria for Adverse Events Scale Version 2.0, Functional Independence Measure Scale, European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 Scale and Visual Analogue Scale for pain before treatment and in 5 weeks of follow-up after treatment.

ELIGIBILITY:
Inclusion Criteria:

Cancer adult patients with CIPN -

Exclusion Criteria:

Other neuropathy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
neurological symptoms | up to 7 weeks
  This study aims to determine the effectiveness of the use of acupuncture in relieving sensory and motor symptoms of patients with chemotherapy induced peripheral neuropathy

SECONDARY OUTCOMES:
functional impairment | up to 7 weeks
  This study aims to determine the effectiveness of the use of acupuncture in relieving functional impairments of patients with chemotherapy induced peripheral neuropathy
quality of life | up to 7 weeks
  This study aims to determine the influence of the use of acupuncture in quality of life of patients with chemotherapy induced peripheral neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca B Cecatto, PhD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Cancer do Estado de São Paulo ICESP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] D'Alessandro EG, Nebuloni Nagy DR, de Brito CMM, Almeida EPM, Battistella LR, Cecatto RB. Acupuncture for chemotherapy-induced peripheral neuropathy: a randomised controlled pilot study. BMJ Support Palliat Care. 2022 Mar;12(1):64-72. doi: 10.1136/bmjspcare-2018-001542. Epub 2019 Jun 29. PMID 31256014